CLINICAL TRIAL: NCT00959465
Title: An Open Label Phase 1/2 Study to Assess Immunogenicity and Safety of Different Dose Levels of H1N1 Pandemic Influenza Vaccine in Healthy Adults Aged 18 Years and Older
Brief Title: A/H1N1 Immunogenicity and Safety in Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Gerald Aichinger, MD; Study Medical Director, Baxter Healthcare Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 820902; EUDRACT Number 2009-013394-17
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2010-07

CONDITIONS: Influenza; Pandemic Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1/Dose Level A (Experimental): Subjects in Cohort 1 will be randomized 1:1 to receive two vaccinations of Dose A or Dose B of H1N1 pandemic influenza vaccine at a 21-day interval.
  Interventions: Biological: H1N1 pandemic influenza vaccine (whole virion, Vero Cell-derived, inactivated)
- Cohort 1/Dose B (Experimental): Subjects in Cohort 1 will be randomized 1:1 to receive two vaccinations of Dose A or Dose B of H1N1 pandemic influenza vaccine at a 21-day interval.
  Interventions: Biological: H1N1 pandemic influenza vaccine (whole virion, Vero Cell-derived, inactivated)
- Cohort 2/Dose C (Experimental): A second cohort may be enrolled with all subjects in this cohort receiving two vaccinations of Dose C of H1N1 pandemic influenza vaccine at a 21-day interval.
  Interventions: Biological: H1N1 pandemic influenza vaccine (whole virion, Vero Cell-derived, inactivated)

INTERVENTIONS:
Biological: H1N1 pandemic influenza vaccine (whole virion, Vero Cell-derived, inactivated) — Two injections at a 21-day interval (Days 1 and 22)

SUMMARY:
The purpose of the study is to obtain immunogenicity and safety data at different dose levels of an investigational H1N1 pandemic influenza vaccine in healthy adults 18 years of age and older.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 to 59 years old (age stratum A) or 60 years of age or older (age stratum B) at the time of screening
* Subject has an understanding of the study, agrees to its provisions, and gives written informed consent prior to study entry
* Subject is generally healthy, as determined by the investigator's clinical judgment through collection of medical history and the performance of a physical examination
* Subject is physically and mentally capable of participating in the study and willing to adhere to study procedures to include completion of all elements of the study diary
* If female of childbearing potential, subject has a negative urine pregnancy test result within 24 hours prior to the scheduled first vaccination and agrees to employ adequate birth control measures for the duration of the study

Exclusion Criteria:

* Subject has participated in another clinical study involving an investigational drug, biological product or device within 30 days prior to study enrollment or is scheduled to participate in another clinical study involving an investigational drug, biological or device during the course of this study
* Subject has a history of exposure to A/H1N1/California/07/2009 virus or a history of vaccination with A/H1N1/California/07/2009 antigen or a closely related influenza virus antigen
* Subject has inherited or acquired immune deficiency
* Subject currently has or has a recent history of significant neurological, cardiovascular or pulmonary (including asthma), hepatic, metabolic, rheumatic, autoimmune, hematological or renal disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2009-08; Primary Completion 2009-11 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Number of subjects achieving antibody levels to A/H1N1/California/07/2009 virus that meet the definition of seroprotection and seroconversion at 21 days after the second vaccination | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Aichinger, MD, Study Director — Baxter Healthcare Corporation
Locations (5):
- Austria (4):
  - Sanatorium Leech, Graz
  - ClinPharm International GmbH, Vienna
  - Medical University of Vienna, Institute for Specific Prophylaxis and Tropical Medicine, Vienna
  - University Hospital, Department of Clinical Pharmacology, Vienna
- Praxis Regner Schmitt, Mainz, Germany